CLINICAL TRIAL: NCT01125618
Title: A Pair-matched Community Intervention Trial to Assess the Impact of an Integrated Health and Development Intervention on Child Survival and the Millennium Development Goals in 10 Sub- Saharan African Countries
Brief Title: Millennium Villages Project in Sub-Saharan Africa
Acronym: MVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United Nations (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Sonia Sachs, Director of Health, The Earth Institute, Columbia University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AAAA8202
Record Dates: First submitted 2010-05-12; First posted 2010-05-18 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Child Survival
Keywords: child mortality; intervention; Poverty; Africa; Millennium Development Goal; Millennium Development Goals
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVP village (Experimental): Wealth stratified and randomly selected households residing in a village exposed to the Millennium Villages Project intervention (or health and development intervention package)
  Interventions: Other: Health and development intervention package
- Comparison village (Active Comparator): Villages receiving routine services through established programs
  Interventions: Other: Routine services

INTERVENTIONS:
Other: Health and development intervention package — The timing and sequence of intervention vary by site, but include improved access to seed-fertilizer to increase agricultural production; improved market and capital access; proven maternal-newborn-child health interventions delivered free of cost at the point of service; improvements to school number and quality; and access to basic infrastructure including safe water, sanitation, electricity, transport and communication.
  Other Names: maternal-newborn-child health interventions; MVP
  Arms: MVP village
Other: Routine services — Routine services and programs currently being administered using prevailing resources, at the current pace and with established partnerships. There is no attempt to limit the introduction of new interventions or agencies into comparison sites.
  Other Names: standard of care services
  Arms: Comparison village

SUMMARY:
The Millennium Villages Project involves the coordinated and simultaneous delivery of a package of proven interventions in health, agriculture, infrastructure and education. The project works in partnership with governments in 10 African countries in areas where progress towards achieving the Millennium Development Goals has been insufficient.

The Project evaluation will test the following hypotheses:

1. That after 5 years of operation, villages exposed to the MVP intervention will have a lower rate of under-5 mortality and parallel gains in MDG-related secondary outcomes when compared to similar villages not receiving the intervention.
2. That the coordinated delivery a multi-sector package of health and development interventions implemented through a broad-based local partnership is feasible in a diversity of sub-Saharan African contexts, and;
3. The intervention package can be delivered at a scalable cost of $40 per person per year in the health sector and $110 per person per year in total

DETAILED DESCRIPTION:
Design and population The design is a pair-matched community intervention trial. Village clusters with high levels of malnutrition were selected from rural areas in ten sub-Saharan African countries to reflect a diverse range of agro-ecological zones, farming systems, disease profiles, and infrastructure challenges. MVP sites represent 80 villages in 14 clusters across 10 countries, covering nearly 500,000 people. For each intervention cluster, a matched comparison cluster has been selected at random to participate in the evaluation.

Outcomes The primary outcome is the under-5 mortality rate. Secondary outcomes are levels of coverage with essential maternal-child health interventions and related MDG indicators for poverty, nutrition, education, and environmental health.

Sample size calculation The assessment follows 6000 households across intervention and matched comparison villages at baseline, and after 3 and 5 years of intervention exposure. With 10 paired clusters, the study is powered to detect a 40% difference in the U5MR between the two groups.

Analysis plan The analysis will use a two-staged pair-matched cluster level analysis, and will be complemented with multilevel modeling. Reporting will adhere to Transparent Reporting of Evaluations with Non-randomized Designs (TREND) guidelines.

Implementation science A portfolio of qualitative implementation science (process evaluation) will complement the quantitative assessment, and involves interviews with implementers, partners, and project beneficiaries. This analysis will address questions about: the feasibility of the interventions; the timing and sequence of their introduction; key contextual barriers and facilitators to implementation; and potential synergies achieved from the integrated multisector approach.

Economic costing study One project hypothesis is that an annual per capita investment of $110 is required to achieve the MDGs. The aim of the economic costing study is to document the absolute and relative contribution of project partners (MVP, government, donors, and the community) to all priced and non-priced cluster-level activities, as well as the sector-specific breakdown of these inputs.

ELIGIBILITY:
Inclusion Criteria:

* Resident in a Millennium Village and consenting to periodic assessments

Exclusion Criteria:

* Those not consenting to participate

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65000 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2016-06-25 (Actual); Study Completion 2016-06-25 (Actual)

PRIMARY OUTCOMES:
Child Mortality Rate | 5 years
  Under 5 Mortality Rate

SECONDARY OUTCOMES:
Prevalence of Stunting | 5 years
  Proportion of under 5s who are stunted; Stunted = low height for age Z-score
Prevalence of Diarrhea | 5 years
  Proportion of under 5's with diarrhea in past 2 weeks
Prevalence of Malaria | 5 years
  Prevalence of malaria among under 5s at the time of survey
Prevalence of antenatal care | 5 years
  Proportion of women who receive at least 4 ANC visits
Survival rate to last grade of primary education (School Quality) | 5 years
Prevalence of improved sanitation utilization | 5 years
  Proportion of the population using an improved sanitation source
Duration or breast feeding (Child feeding practices) | 5 years
Age of introduction of complementary feeding (Child feeding practices) | 5 years
Prevalence of bed net utilization | 5 years
  Proportion of under 5s sleeping under Longlasting insecticide treated bednets in the night prior to the survey
Prevalence of malaria treatment | 5 years
  Proportion of under 5s with a fever in the past 2 weeks who receive appropriate anti-malarial treatment
Prevalence of measles immunization | 5 years
  Proportion under 1s immunized against measles
Prevalence of diarrhea management | 5 years
  Proportion of under 5s with diarrhea in the past 2 weeks who received oral rehydration therapy
Prevalence of pneumonia management | 5 years
  Proportion of under 5s treated for pneumonia in the past 2 weeks
Prevalence of newborn care | 5 years
  Proportion of newborns receiving a post-natal check in the first week of life
Proportion of pregnant women who received and HIV test | 5 years
  This measures the prevention of vertical transmission of HIV
Prevalence of food insecurity | 5 years
  Proportion of households reporting not enough food for 1 of past 12 months
Institutional delivery rate | 5 years
  Proportion of births attended by skilled health personnel
Prevalence of underweight | 5 years
  Proportion of under 5s who are underweight; Underweight= weight for age Z score
Prevalence of wasting | 5 years
  Proportion of under 5s who are wasted; Wasting = weight for height Z score
Prevalence of low mid-upper arm circumference | 5 years
  Proportion of under 5s with a low mid-upper arm circumference
Household Asset Index (Household poverty) | 5 years
  Survey of fixed and non-fixed assets, including recent purchases
Prevalence of improved water source utilization | 5 years
  Proportion of the population using an improved drinking water source

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sachs, PhD, Study Chair — The Earth Institute, Columbia University; Pedro Sanchez, PhD, Study Director — The Earth Institute, Columbia University; Cheryl Palm, PhD, Principal Investigator — The Earth Institute, Columbia University; Sonia Sachs, MD, PhD, Principal Investigator — Director of Health, The Earth Institute, Columbia University
Locations (11):
- Koraro, Koraro, Ethiopia
- Bonsasso, Bonsasso, Ghana
- Sauri, Sauri, Kenya
- Mwandama, Mwandama, Malawi
- Tiby, Tiby, Mali
- Nigeria (2):
  - Ikaram, Ikaram
  - Pampaida, Pampaida
- Mayange, Mayange, Rwanda
- Potou, Potou, Senegal
- Mbola, Mbola, Tanzania
- Ruhiira, Ruhiira, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pronyk PM, Muniz M, Nemser B, Somers MA, McClellan L, Palm CA, Huynh UK, Ben Amor Y, Begashaw B, McArthur JW, Niang A, Sachs SE, Singh P, Teklehaimanot A, Sachs JD; Millennium Villages Study Group. The effect of an integrated multisector model for achieving the Millennium Development Goals and improving child survival in rural sub-Saharan Africa: a non-randomised controlled assessment. Lancet. 2012 Jun 9;379(9832):2179-88. doi: 10.1016/S0140-6736(12)60207-4. Epub 2012 May 8. PMID 22572602